CLINICAL TRIAL: NCT05526131
Title: Brain Derived Neurotropic Factor Level and val66met Polymorphism of Brain Derived Neurotropic Factor Gene in Patients With Type Two Diabetes Mellitus and Depression
Brief Title: BDNF Level and val66met Polymorphism of Brain Derived Neurotropic Factor Gene in Patients With T2DM and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Tarek Samy Abdelaziz, Associate professor, Kasr El Aini Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: KA-239-D
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Depression; Diabetes Mellitus
Keywords: Brain Derived Neurotrophic Factor; Diabetes Mellitus
MeSH Terms: conditions — Depression; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with type 2 Diabetes Mellitus and depression (Active Comparator): This arm includes patients with type 2 diabetes mellitus that were diagnosed with depression using structured clinical interview for DSM-IV Axis disorder (SCID-I) and Hamilton Depression Rating Scale (HAM-D) for diagnosing depression and exclusion of other psychiatric disorders.
  Interventions: Other: Questionare
- Patients with type 2 Diabetes Mellitus and no depression (Active Comparator): This arm includes patients with type 2 diabetes mellitus where depression was ruled out using structured clinical interview for DSM-IV Axis disorder (SCID-I) and Hamilton Depression Rating Scale (HAM-D) for diagnosing depression and exclusion of other psychiatric disorders.
  Interventions: Other: Questionare

INTERVENTIONS:
Other: Questionare — Assessing the presence or the absence of depression:
  By structured clinical interview for DSM-IV Axis disorder (SCID-I) and Hamilton Depression Rating Scale (HAM-D) for diagnosing depression and exclusion of other psychiatric disorders.

SUMMARY:
This study aimed to evaluate the relation between the levels of (Brain Derived Neurotropic Factor) BDNF and val66met polymorphism of BDNF gene, and the presence of depression in type 2 diabetes. In addition to studying the relationship between BDNF level and val66met polymorphism of its gene and assessing relation between BDNF level and obesity.

DETAILED DESCRIPTION:
The study included 88 type 2 diabetic patients, which are further divided into two groups; depressed and non-depressed. Depression was assessed by Hamilton Depression Rating Scale (HAM-D) and structured clinical interview for DSM-IV Axis disorder (SCID-I) for diagnosing depression and exclusion of other psychiatric disorders. Genotyping was performed by using Real Time-PCR (TaqMan probes).

ELIGIBILITY:
Adult patients who have type two diabetes with or without depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-10-23 (Actual)

PRIMARY OUTCOMES:
BDNF level in blood | 1 day (At the time of recruitment)
  Measurement of the level of BDNF in blood
val66met polymorphism of BDNF gene | 1 day (At the time of recruitment)
  Measurement of val66met polymorphism of BDNF gene

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Abdelaziz, PhD, Principal Investigator — Kasr Alaini University Hsopitals
Locations (1):
- Cairo university hospitals, Cairo, Egypt